CLINICAL TRIAL: NCT04504656
Title: Comparison of Early Outcomes of Minimally Invasive Surgery for Oesophageal Replacement Versus Open Surgery in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A maher, Assistant lecturer of surgery, Assiut University
Other Study IDs: Esophageal replacement
Record Dates: First submitted 2020-08-01; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Post-Op Complication; Anastomosis; Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Constriction; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: open surgery
  Interventions: Other: observation of postoperative leak, stenosis, mortality
- 2: minimally invasive surgery
  Interventions: Other: observation of postoperative leak, stenosis, mortality

INTERVENTIONS:
Other: observation of postoperative leak, stenosis, mortality — detect complications in both groups

SUMMARY:
a comparative prospective study of postoperative between minimally invasive and open surgery complications for esophageal replacement in children

DETAILED DESCRIPTION:
Esophageal replacement in childhood is indicated in esophageal atresia patients with long-gap defects or following complications of primary esophageal anastomosis, as well as in patients with trauma and scarring to the esophagus following caustic ingestion. It is widely accepted that the ideal esophageal replacement is one that resembles the function of the native esophagus with minimal deterioration over time. Several techniques of esophageal replacement have been developed. These have focused mainly on the use of native tissues (including the stomach, jejunum, and colon) as conduits (1), attempts to use a synthetic prosthesis have been largely unsuccessful. In an attempt to reduce the trauma and morbidity associated with laparotomy and thoracotomy incisions, minimally invasive techniques are increasingly used. (2-4). Meta-analyses of adult esophagectomy for the treatment of esophageal cancer support the use of minimally invasive surgery (5) however, equivalent comparative studies in the pediatric population are lacking. As such, it is unclear whether minimally esophageal replacement is as safe as the open procedure in children. The present study aims to address this question by comparing the postoperative outcomes of children who underwent minimally invasive versus open esophageal replacement procedures at single-center and multicenter levels.

ELIGIBILITY:
Inclusion Criteria:

All children undergoing oesophageal replacement aged one to 18 years. Due to

1. long gap esophageal atresia
2. caustic ingestion
3. congenital esophageal stenosis or strictures

Exclusion Criteria:

* patient who underwent previous esophageal replacement operations.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children up to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Anastamotic leaks | 2 years
  Incidence of anastamotic leak which is identified clinically in both groups

SECONDARY OUTCOMES:
Anastamotic stricture | 2 years
  Incidence of symptomstic strictures which is identified by upper barium studies
Mortality | 2 years
  Number of patient who die intraoperative and post operative in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Eltayeb, MD, Study Director — Assiut University
Locations (1):
- Assiut University Children Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol